CLINICAL TRIAL: NCT03979872
Title: Risk Information and Skin-cancer Education for Undergraduate Prevention
Acronym: RISE-UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Yelena Wu, Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB_00116807
Record Dates: First submitted 2019-06-05; First posted 2019-06-07 (Actual); Results first posted 2021-07-01 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Melanoma; Young Adult
Keywords: Education Prevention; MC1R Genetic Testing
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: 4 different parallel intervention groups:
  * Education only
  * Education + MC1R genetic testing
  * Education + UV photo
  * Education + MC1R genetic testing + UV photo
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1: Skin Cancer Education Only (Active Comparator): Participants will be randomized to receive education only.
  Interventions: Other: Skin Cancer Education
- Arm 2: Skin Cancer Education + UV Photo (Experimental): Participants randomized to receive education + UV photo will have a UV light photo taken of their face to show UV damage in the skin that is invisible to the naked eye in addition to receiving skin cancer education.
  Interventions: Other: Skin Cancer Education; Device: UV Photo
- Arm 3: Skin Cancer Education + MC1R Testing (Experimental): Participants randomized to receive education + genetic testing will be asked to provide a saliva sample for MC1R testing in addition to receiving skin cancer education.
  Interventions: Diagnostic Test: MC1R Genetic Testing; Other: Skin Cancer Education
- Arm 4: Skin Cancer Education + UV Photo + MC1R Testing (Experimental): Participants randomized to receive education + UV photo + genetic testing will have a UV light photo taken of their face, Submit a saliva sample for MC1R testing, and receive skin cancer education.
  Interventions: Diagnostic Test: MC1R Genetic Testing; Other: Skin Cancer Education; Device: UV Photo

INTERVENTIONS:
Diagnostic Test: MC1R Genetic Testing — [See arm/group descriptions]
  Arms: Arm 3: Skin Cancer Education + MC1R Testing; Arm 4: Skin Cancer Education + UV Photo + MC1R Testing
Other: Skin Cancer Education — [See arm/group descriptions]
Device: UV Photo — [See arm/group descriptions]
  Arms: Arm 2: Skin Cancer Education + UV Photo; Arm 4: Skin Cancer Education + UV Photo + MC1R Testing

SUMMARY:
The purpose of this study will be to provide undergraduate students information about skin cancer risk and prevention. The study will last between 2-3 months. Everyone in the study will be asked to answer questionnaires and receive education about skin cancer risk factors and prevention. We will follow-up with participants by phone, text messages or e-mail in between study visits

Participants will be randomly assigned to one of four groups, the group will be in is decided by chance. Participant will either be assigned to:

* A group that gets advice about what causes skin cancer and how to prevent it
* A group that gets this advice and provides a saliva sample to receive personalized skin cancer risk genetic testing results
* A group that gets this advice and receives a personalized photo that shows existing skin damage
* A group that gets this advice, receives genetic testing results, and receives a personalized photo.

DETAILED DESCRIPTION:
Arm 1: Skin Cancer Education Only

Screening: Participants will have the option to complete and online or text based screening form. Study staff may contact participants who screen to be eligible via phone, text, or email. Study staff will screen potential participants who do not complete the screening form on their own for eligibility. Participants will be contacted by phone, text, or email (starting with the method they indicated would be best to reach them) to schedule their first study visit.

Enrollment

Visit 1: All participants who consent to participate will be asked to participate in up to 3 study visits approximately 4 weeks apart. At visit 1, all participants will be asked to complete informed consent procedures and a baseline questionnaire via computer (e.g., using Qualtrics) or paper. Participants will be randomized to receive education only, or varying combinations of the intervention components.

Visit 2: At visit 2 participants will receive education on the importance of skin cancer prevention behaviors (e.g., sunscreen, protective clothing) and avoiding tanning and sunburns. All education will be delivered at this visit on a computer screen and additionally given to participants as a handout they can take home to review. When participants view the information on the computer screen, eye tracking will be used to assess participant response. Prior to viewing results, eye tracking equipment set up at the computer station will be calibrated. We will then put up their results on the screen and the imotion system will then track their pupillary movement, facial expression, and galvanic skin response (physiological arousal). Participants will be allowed as much time as they would like to review their results. Following this, participants will complete a post assessment. Participants will receive paper copies of all of the relevant information to take home with them.

Visit 3: Visit 3 may be conducted remotely. At visit 3, participants will complete a follow-up assessment.

Follow-up interview: A random sample of the participant population with be contacted to participate in a follow-up interview with study staff to answer questions about their experience participating in the RISE-UP study.

Arm 2: Skin Cancer Education + UV Photo

Screening: Participants will have the option to complete and online or text based screening form. Study staff may contact participants who screen to be eligible via phone, text, or email.Study staff will screen potential participants who do not complete the screening form on their own for eligibility. Participants will be contacted by phone, text, or email (starting with the method they indicated would be best to reach them) to schedule their first study visit.

Enrollment

Visit 1: All participants who consent to participate will be asked to participate in up to 3 study visits approximately 4 weeks apart. At visit 1, all participants will be asked to complete informed consent procedures and a baseline questionnaire via computer (e.g., using Qualtrics) or paper. Participants will be randomized to receive education only, or varying combinations of the intervention components. Participants randomized to the education + UV photo arm will have their UV light photo taken of their face to show UV damage in the skin that is invisible to the naked eye. Photos will be taken with the VISIA Facial Complexion Analysis System, which captures high resolution imagery at the far spectrum of UVA or long wave UV.

Visit 2: At visit 2 participants will receive education on the importance of skin cancer prevention behaviors (e.g., sunscreen, protective clothing) and avoiding tanning and sunburns. Participants will be provided with their personalized risk feedback based on their personalized photo showing their skin's existing UVR damage from UVR exposure. All information will be delivered at this visit on a computer screen and additionally given to participants as a handout they can take home to review. When participants view their results on the computer screen, eye tracking will be used to assess participant response. Prior to viewing results, eye tracking equipment set up at the computer station will be calibrated. We will then put up their results on the screen and the imotion system will then track their pupillary movement, facial expression, and galvanic skin response (physiological arousal). Participants will be allowed as much time as they would like to review their results. Following this, participants will complete a post assessment. The imagery resulting will be kept on file in a password protected computer. Participants will receive paper copies of all of the relevant information to take home with them.

Visit 3: Visit 3 may be conducted remotely. At visit 3, participants will complete a follow-up assessment.

Follow-up interview: A random sample of the participant population with be contacted to participate in a follow-up interview with study staff to answer questions about their experience participating in the RISE-UP study.

Arm 3: Skin Cancer Education + MC1R Testing

Screening: Participants will have the option to complete and online or text based screening form. Study staff may contact participants who screen to be eligible via phone, text, or email.Study staff will screen potential participants who do not complete the screening form on their own for eligibility. Participants will be contacted by phone, text, or email (starting with the method they indicated would be best to reach them) to schedule their first study visit.

Enrollment

Visit 1: All participants who consent to participate will be asked to participate in up to 3 study visits approximately 4 weeks apart. At visit 1, all participants will be asked to complete informed consent procedures and a baseline questionnaire via computer (e.g., using Qualtrics) or paper. Participants will be randomized to receive education only, or varying combinations of the intervention components. Participants randomized to the education + MC1R testing arm will be asked to be provide a saliva sample. Saliva will be collected by study staff using a system for the collection, stabilization and transportation of DNA from saliva (e.g., Oragene DNA collection kits). Molecular evaluation will be performed at the genetic, enzymatic (protein and RNA), and cellular response levels to identify melanoma predisposition genes.

Visit 2: At visit 2 participants will receive education on the importance of skin cancer prevention behaviors (e.g., sunscreen, protective clothing) and avoiding tanning and sunburns. Participants will be provided with their personalized risk feedback based on a summary of their MC1R genetic testing results. All information will be delivered at this visit on a computer screen and additionally given to participants as a handout they can take home to review. When participants view their results on the computer screen, eye tracking will be used to assess participant response. Prior to viewing results, eye tracking equipment set up at the computer station will be calibrated. We will then put up their results on the screen and the imotion system will then track their pupillary movement, facial expression, and galvanic skin response (physiological arousal). Participants will be allowed as much time as they would like to review their results. Following this, participants will complete a post assessment. Participants will receive paper copies of all of the relevant information to take home with them.

Visit 3: Visit 3 may be conducted remotely. At visit 3, participants will complete a follow-up assessment. After visit 3, participants will be offered the option to opt-in to receiving their raw genetic test report.

Follow-up interview: A random sample of the participant population with be contacted to participate in a follow-up interview with study staff to answer questions about their experience participating in the RISE-UP study.

Arm 4: Skin Cancer Education + UV Photo + MC1R Testing

Screening: Participants will have the option to complete and online or text based screening form. Study staff may contact participants who screen to be eligible via phone, text, or email.Study staff will screen potential participants who do not complete the screening form on their own for eligibility. Participants will be contacted by phone, text, or email (starting with the method they indicated would be best to reach them) to schedule their first study visit.

Enrollment

Visit 1: All participants who consent to participate will be asked to participate in up to 3 study visits approximately 4 weeks apart. At visit 1, all participants will be asked to complete informed consent procedures and a baseline questionnaire via computer (e.g., using Qualtrics) or paper. Participants will be randomized to receive education only, or varying combinations of the intervention components. Participants randomized to the education + UV photo + MC1R testing arm will have a UV light photo taken of their face to show UV damage in the skin that is invisible to the naked eye and will be asked to provide a saliva sample. Photos will be taken with the VISIA Facial Complexion Analysis System, which captures high resolution imagery at the far spectrum of UVA or long wave UV. Saliva will be collected by study staff using a system for the collection, stabilization and transportation of DNA from saliva (e.g., Oragene DNA collection kits). Molecular evaluation will be performed at the genetic, enzymatic (protein and RNA), and cellular response levels to identify melanoma predisposition genes.

Visit 2: At visit 2 participants will receive education on the importance of skin cancer prevention behaviors (e.g., sunscreen, protective clothing) and avoiding tanning and sunburns. Participants will be provided with their personalized risk feedback based on a summary of their personalize UV photo and a summary of their MC1R genetic testing results. All information will be delivered at this visit on a computer screen and additionally given to participants as a handout they can take home to review. When participants view their results on the computer screen, eye tracking will be used to assess participant response. Prior to viewing results, eye tracking equipment set up at the computer station will be calibrated. We will then put up their results on the screen and the imotion system will then track their pupillary movement, facial expression, and galvanic skin response (physiological arousal). Participants will be allowed as much time as they would like to review their results. Following this, participants will complete a post assessment. The imagery resulting will be kept on file in a password protected computer. Participants will receive paper copies of all of the relevant information to take home with them.

Visit 3: Visit 3 may be conducted remotely. At visit 3, participants will complete a follow-up assessment. After visit 3, participants will be offered the option to opt-in to receiving their raw genetic test report.

Follow-up interview: A random sample of the participant population with be contacted to participate in a follow-up interview with study staff to answer questions about their experience participating in the RISE-UP study.

ELIGIBILITY:
Inclusion Criteria:

* Individual is enrolled in courses at the University of Utah

And

* Individual reports having had at least 1 sunburn in the past year

And/or

* Individual reports having intentionally indoor or outdoor tanned at lease 1 time in the past year

And/or

- Individual reports using sunscreen plus 1 or more other following behaviors never/rarely/sometimes in the past month: 1)Protective clothing items, 2)Shade when outdoors

Exclusion Criteria:

* Individual does not read/speak English
* Individual reports a personal history of skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2020-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yelena Wu, PHD, Principal Investigator — University of Utah
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Wu YP, Hamilton JG, Kaphingst KA, Jensen JD, Kohlmann W, Parsons BG, Lillie HM, Wang X, Haaland B, Wankier AP, Grossman D, Hay JL. Increasing Skin Cancer Prevention in Young Adults: the Cumulative Impact of Personalized UV Photography and MC1R Genetic Testing. J Cancer Educ. 2023 Jun;38(3):1059-1065. doi: 10.1007/s13187-022-02232-1. Epub 2022 Oct 28. PMID 36306029

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Students were recruited from a 4-year public university
Period: Overall Study
Arm/Group | Arm 1: Skin Cancer Education Only | Arm 2: Skin Cancer Education + UV Photo | Arm 3: Skin Cancer Education + MC1R Testing | Arm 4: Skin Cancer Education + UV Photo + MC1R Testing
Started | 22 | 23 | 24 | 23
Completed | 19 | 15 | 18 | 19
Not Completed | 3 | 8 | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Skin Cancer Education Only | Arm 2: Skin Cancer Education + UV Photo | Arm 3: Skin Cancer Education + MC1R Testing | Arm 4: Skin Cancer Education + UV Photo + MC1R Testing | Total
Number analyzed (Participants) | 22 | 23 | 24 | 23 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 23 | 24 | 23 | 92
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 17 | 16 | 65
  Male | 6 | 7 | 7 | 7 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 2 | 2 | 7
  Not Hispanic or Latino | 16 | 18 | 19 | 12 | 65
  Unknown or Not Reported | 3 | 5 | 3 | 9 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 17 | 18 | 21 | 14 | 70
  More than one race | 5 | 4 | 0 | 3 | 12
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 22 | 23 | 24 | 23 | 92

OUTCOME MEASURES:

1. Primary Outcome: Sun Protection Behaviors Assessed Via Questionnaires
Description: Mean and standard deviation for each sun protection behavior at Visit 1 (baseline), Visit 2 (4 weeks), Visit 3 (8 weeks).
  "These next questions ask about what you have done in the past four weeks if you were outdoors in the sun for 15 minutes or more. How often did you... " Minimum value =1; Maximum value= 5; Higher scores indicate that participants were more likely to engage in sun protection habits.
Time Frame: Weeks 0 (Visit 1), 4 (Visit 2), 8 (Visit 3)
Population: The difference in the number of participants analyzed at each visit versus overall participants analyzed for each study arm is due to participant attrition over time.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Skin Cancer Education Only | Arm 2: Skin Cancer Education + UV Photo | Arm 3: Skin Cancer Education + MC1R Testing | Arm 4: Skin Cancer Education + UV Photo + MC1R Testing
Number analyzed (Participants) | 22 | 23 | 24 | 23
score on a scale
  Sun Protection- Sunscreen Visit 1 | 2.4 (1.2) | 3.0 (1.2) | 2.8 (1.3) | 2.3 (1.1)
  Sun Protection- Sunscreen Visit 2: number analyzed (Participants) | 20 | 20 | 22 | 22
  Sun Protection- Sunscreen Visit 2 | 2.4 (1.0) | 2.4 (1.4) | 2.7 (1.4) | 2.1 (1.2)
  Sun Protection- Sunscreen Visit 3: number analyzed (Participants) | 19 | 15 | 18 | 19
  Sun Protection- Sunscreen Visit 3 | 2.3 (1.3) | 2.9 (1.2) | 2.3 (1.6) | 2.2 (1.1)
  Sun Protection- Reapply sunscreen Visit 1 | 1.6 (1.0) | 1.9 (1.0) | 2.0 (1.1) | 1.9 (0.8)
  Sun Protection- Reapply sunscreen Visit 2: number analyzed (Participants) | 20 | 20 | 22 | 22
  Sun Protection- Reapply sunscreen Visit 2 | 1.6 (1.1) | 1.6 (0.9) | 1.8 (1.1) | 1.3 (0.6)
  Sun Protection- Reapply sunscreen Visit 3: number analyzed (Participants) | 19 | 15 | 18 | 19
  Sun Protection- Reapply sunscreen Visit 3 | 2.2 (1.1) | 1.5 (1.0) | 1.7 (1.1) | 1.6 (1.0)
  Sun Protection- Shirt with sleeves Visit 1 | 3.9 (1.1) | 4.0 (0.9) | 4.0 (0.9) | 3.6 (1.5)
  Sun Protection- Shirt with sleeves Visit 2: number analyzed (Participants) | 20 | 20 | 22 | 22
  Sun Protection- Shirt with sleeves Visit 2 | 3.8 (1.2) | 3.9 (1.5) | 4.1 (1.1) | 4.1 (1.0)
  Sun Protection- Shirt with sleeves Visit 3: number analyzed (Participants) | 19 | 15 | 18 | 19
  Sun Protection- Shirt with sleeves Visit 3 | 3.9 (1.1) | 4.5 (0.9) | 3.9 (1.3) | 4.2 (0.9)
  Sun Protection- Long pants/long skirt Visit 1 | 3.4 (1.1) | 3.3 (1.2) | 3.6 (1.2) | 3.6 (1.5)
  Sun Protection- Long pants/long skirt Visit 2: number analyzed (Participants) | 20 | 20 | 22 | 22
  Sun Protection- Long pants/long skirt Visit 2 | 3.6 (1.2) | 3.5 (1.6) | 3.9 (1.3) | 4.1 (1.0)
  Sun Protection- Long pants/long skirt Visit 3: number analyzed (Participants) | 19 | 15 | 18 | 19
  Sun Protection- Long pants/long skirt Visit 3 | 3.7 (1.1) | 4.0 (1.1) | 4.1 (1.1) | 4.1 (1.0)
  Sun Protection- Hat Visit 1 | 1.9 (0.9) | 1.9 (1.2) | 1.6 (0.8) | 1.2 (0.4)
  Sun Protection- Hat Visit 2: number analyzed (Participants) | 20 | 20 | 22 | 22
  Sun Protection- Hat Visit 2 | 1.9 (1.0) | 1.9 (1.3) | 1.8 (1.0) | 1.4 (0.9)
  Sun Protection- Hat Visit 3: number analyzed (Participants) | 19 | 15 | 18 | 19
  Sun Protection- Hat Visit 3 | 1.8 (0.8) | 1.9 (1.3) | 1.3 (0.6) | 1.4 (0.5)
  Sun Protection- Shade or Umbrella Visit 1 | 2.3 (1.0) | 2.8 (1.1) | 2.6 (0.9) | 2.5 (0.8)
  Sun Protection- Shade or Umbrella Visit 2: number analyzed (Participants) | 20 | 20 | 22 | 22
  Sun Protection- Shade or Umbrella Visit 2 | 2.4 (1.3) | 3.0 (1.4) | 2.1 (1.1) | 2.5 (1.1)
  Sun Protection- Shade or Umbrella Visit 3: number analyzed (Participants) | 19 | 15 | 18 | 19
  Sun Protection- Shade or Umbrella Visit 3 | 2.6 (1.0) | 2.9 (1.2) | 2.4 (1.3) | 2.9 (1.2)
  Sun Protection- Avoid sun during peak hours Visit 1 | 2.1 (1.0) | 2.4 (1.1) | 2.1 (0.9) | 2.0 (0.9)
  Sun Protection- Avoid sun during peak hours Visit 2: number analyzed (Participants) | 20 | 20 | 22 | 22
  Sun Protection- Avoid sun during peak hours Visit 2 | 2.1 (1.1) | 2.4 (1.3) | 2.2 (1.1) | 2.6 (1.0)
  Sun Protection- Avoid sun during peak hours Visit 3: number analyzed (Participants) | 19 | 15 | 18 | 19
  Sun Protection- Avoid sun during peak hours Visit 3 | 2.5 (1.1) | 3.0 (1.0) | 2.6 (1.2) | 2.8 (1.0)
  Sun Protection- Sunglasses Visit 1 | 3.0 (1.1) | 2.6 (1.4) | 2.8 (1.2) | 2.8 (1.4)
  Sun Protection- Sunglasses Visit 2: number analyzed (Participants) | 20 | 20 | 22 | 22
  Sun Protection- Sunglasses Visit 2 | 2.1 (1.1) | 2.7 (1.6) | 3.1 (1.3) | 2.5 (1.5)
  Sun Protection- Sunglasses Visit 3: number analyzed (Participants) | 19 | 15 | 18 | 19
  Sun Protection- Sunglasses Visit 3 | 2.5 (1.1) | 2.5 (1.8) | 2.9 (1.1) | 2.1 (1.3)

2. Secondary Outcome: Sunburn Occurrence Assessed Via Questionnaire
Description: Average number of sunburns received by participants in the past 4 weeks when asked at Visit 1 (baseline), Visit 2 (4 weeks), and Visit 3 (8 weeks)
Time Frame: Weeks 0 (Visit 1), 4 (Visit 2), 8 (Visit 3)
Population: Participants either dropping out or no showing.
Measure: Mean (Standard Deviation); unit: sunburns
Arm/Group | Arm 1: Skin Cancer Education Only | Arm 2: Skin Cancer Education + UV Photo | Arm 3: Skin Cancer Education + MC1R Testing | Arm 4: Skin Cancer Education + UV Photo + MC1R Testing
Number analyzed (Participants) | 22 | 23 | 24 | 23
sunburns
  Visit 1 | 1.14 (.468) | 1.30 (.559) | 1.38 (.875) | 1.13 (.458)
  Visit 2: number analyzed (Participants) | 20 | 20 | 22 | 22
  Visit 2 | 1.50 (1.192) | 1.25 (.716) | 1.23 (.528) | 1.05 (.213)
  Visit 3: number analyzed (Participants) | 19 | 15 | 18 | 23
  Visit 3 | 1.63 (1.300) | 1.67 (1.175) | 1.06 (.236) | 1.16 (.501)

3. Secondary Outcome: Intentional Outdoor Tanning Occurrence Assessed Via Questionnaire
Description: Mean and standard deviation for intentional outdoor tanning occurrences at Visit 1 (baseline), Visit 2 (4 weeks), Visit 3 (8 weeks).
  "In the past 4 Weeks, how often did you spend time in the sun in order to get tan?" Minimum value =1; Maximum value= 5; Higher scores indicates that participants spent more time outdoors to get a tan.
Time Frame: Weeks 0 (Visit 1), 4 (Visit 2), 8 (Visit 3)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Skin Cancer Education Only | Arm 2: Skin Cancer Education + UV Photo | Arm 3: Skin Cancer Education + MC1R Testing | Arm 4: Skin Cancer Education + UV Photo + MC1R Testing
Number analyzed (Participants) | 22 | 23 | 24 | 23
score on a scale
  Visit 1 | 1.8 (1.1) | 1.4 (0.8) | 1.5 (1.1) | 1.6 (0.9)
  Visit 2: number analyzed (Participants) | 20 | 20 | 22 | 22
  Visit 2 | 1.4 (0.8) | 1.2 (0.5) | 1.4 (0.7) | 1.4 (0.9)
  Visit 3: number analyzed (Participants) | 19 | 15 | 18 | 19
  Visit 3 | 1.7 (1.2) | 1.3 (0.8) | 1.1 (0.5) | 1.5 (0.8)

4. Secondary Outcome: Intentional Indoor Tanning Occurrence Assessed Via Questionnaire
Description: Number of times participant used an indoor tanning device in the past 4 weeks when asked at Visit 1 (baseline), Visit 2 (4 weeks), and Visit 3 (8 weeks)
Time Frame: Weeks 0 (Visit 1), 4 (Visit 2), 8 (Visit 3)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Skin Cancer Education Only | Arm 2: Skin Cancer Education + UV Photo | Arm 3: Skin Cancer Education + MC1R Testing | Arm 4: Skin Cancer Education + UV Photo + MC1R Testing
Number analyzed (Participants) | 22 | 23 | 24 | 23
Participants
  Visit 1: 0 times | 22 | 23 | 24 | 23
  Visit 1: 1 or 2 times | 0 | 0 | 0 | 0
  Visit 1: 3 to 9 times | 0 | 0 | 0 | 0
  Visit 1: 10 to 19 times | 0 | 0 | 0 | 0
  Visit 1: 20 to 39 times | 0 | 0 | 0 | 0
  Visit 1: 40 or more times | 0 | 0 | 0 | 0
  Visit 2: number analyzed (Participants) | 20 | 20 | 22 | 22
  Visit 2: 0 times | 19 | 19 | 22 | 21
  Visit 2: 1 or 2 times | 0 | 1 | 0 | 0
  Visit 2: 3 to 9 times | 0 | 0 | 0 | 1
  Visit 2: 10 to 19 times | 1 | 0 | 0 | 0
  Visit 2: 20 to 39 times | 0 | 0 | 0 | 0
  Visit 2: 40 or more times | 0 | 0 | 0 | 0
  Visit 3: number analyzed (Participants) | 19 | 15 | 18 | 19
  Visit 3: 0 times | 17 | 13 | 18 | 17
  Visit 3: 1 or 2 times | 1 | 1 | 0 | 1
  Visit 3: 3 to 9 times | 0 | 1 | 0 | 1
  Visit 3: 10 to 19 times | 1 | 0 | 0 | 0
  Visit 3: 20 to 39 times | 0 | 0 | 0 | 0
  Visit 3: 40 or more times | 0 | 0 | 0 | 0

5. Secondary Outcome: Tan Occurrence Assessed Via Questionnaire
Description: Mean and standard deviation for tan occurrence at Visit 1 (baseline), Visit 2 (4 weeks), Visit 3 (8 weeks).
  "In the past 4 weeks, how often did you end up with a tan, even if you didn't try to get one?" Minimum value =1; Maximum value= 5; Higher scores indicate that participants received a tan as a result or being outdoors or using an indoor tanning device whether intentional or not.
Time Frame: Weeks 0 (Visit 1), 4 (Visit 2), 8 (Visit 3)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Skin Cancer Education Only | Arm 2: Skin Cancer Education + UV Photo | Arm 3: Skin Cancer Education + MC1R Testing | Arm 4: Skin Cancer Education + UV Photo + MC1R Testing
Number analyzed (Participants) | 22 | 23 | 24 | 23
score on a scale
  Visit 1 | 2.3 (1.2) | 2.0 (1.9) | 2.1 (1.3) | 2.0 (1.0)
  Visit 2: number analyzed (Participants) | 20 | 20 | 22 | 22
  Visit 2 | 1.8 (1.1) | 1.6 (1.0) | 1.8 (1.3) | 1.7 (1.0)
  Visit 3: number analyzed (Participants) | 19 | 15 | 18 | 19
  Visit 3 | 1.9 (1.1) | 1.2 (0.6) | 1.2 (0.4) | 1.6 (1.0)

ADVERSE EVENTS:
Time Frame: Each participant was monitored/assessed for adverse events in relation to each visit which occurred every 2 weeks over an 8 week period (a total of 4 times).
Arm/Group | Arm 1: Skin Cancer Education Only | Arm 2: Skin Cancer Education + UV Photo | Arm 3: Skin Cancer Education + MC1R Testing | Arm 4: Skin Cancer Education + UV Photo + MC1R Testing
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/23 | 0/24 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23 | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 0/22 | 0/23 | 0/24 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-24): https://cdn.clinicaltrials.gov/large-docs/72/NCT03979872/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/72/NCT03979872/ICF_001.pdf